CLINICAL TRIAL: NCT05156710
Title: A Multi-cohort, Randomized, Phase 2, Open-label Study to Assess the Preliminary Efficacy, Safety, and Pharmacokinetics of BIVV020 for Prevention and Treatment of Antibody-mediated Rejection in Adult Kidney Transplant Recipients.
Brief Title: BIVV020 (SAR445088) n Prevention and Treatment of Antibody-mediated Rejection (AMR)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT17012; U1111-1267-2612 (Registry Identifier: ICTRP); 2023-509936-25-00 (Registry Identifier: CTIS); 2023-509936-25 (Registry Identifier: CTIS); 2021-000010-41 (EudraCT Number)
Record Dates: First submitted 2021-11-18; First posted 2021-12-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Transplant Rejection
MeSH Terms: interventions — Immunoglobulins, Intravenous; Rituximab; Biosimilar Pharmaceuticals; Antilymphocyte Serum; Tacrolimus; Mycophenolic Acid; Adrenal Cortex Hormones

STUDY DESIGN:
Masking Description: Randomization for Cohort B only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BIVV020 with Standard of Care (SOC) Cohort A (Experimental): Eligible participants will receive BIVV020 and SOC immunosuppression including induction therapy, tacrolimus, and mycophenolate.
  Interventions: Drug: BIVV020 (SAR445088); Drug: Antithymocyte globulin (ATG); Drug: Tacrolimus; Drug: Mycophenolate
- BIVV020 with Standard of Care (SOC) Cohort B (Experimental): Eligible participants will receive BIVV020 and SOC which includes plasmapheresis, IVIg, corticosteroids, rituximab.
  Interventions: Drug: BIVV020 (SAR445088); Drug: Intravenous immunoglobulin (IVIg); Drug: Rituximab or biosimilar; Drug: Corticosteroids
- Standard of Care (SOC) Cohort B (Other): SOC includes plasmapheresis, IVIg, corticosteroids, rituximab.
  Interventions: Drug: Intravenous immunoglobulin (IVIg); Drug: Rituximab or biosimilar; Drug: Corticosteroids

INTERVENTIONS:
Drug: BIVV020 (SAR445088) — Pharmaceutical Form: Solution for injection Route of Administration: Intravenous
  Arms: BIVV020 with Standard of Care (SOC) Cohort A; BIVV020 with Standard of Care (SOC) Cohort B
Drug: Intravenous immunoglobulin (IVIg) — Pharmaceutical Form: Solution for injection Route of Administration: Intravenous
  Arms: BIVV020 with Standard of Care (SOC) Cohort B; Standard of Care (SOC) Cohort B
Drug: Rituximab or biosimilar — Pharmaceutical Form: Solution for injection Route of Administration: Intravenous
  Arms: BIVV020 with Standard of Care (SOC) Cohort B; Standard of Care (SOC) Cohort B
Drug: Antithymocyte globulin (ATG) — Pharmaceutical Form: Solution for injection Route of Administration: Intravenous
  Arms: BIVV020 with Standard of Care (SOC) Cohort A
Drug: Tacrolimus — Pharmaceutical Form: Tablet Route of Administration: Oral
  Arms: BIVV020 with Standard of Care (SOC) Cohort A
Drug: Mycophenolate — Pharmaceutical Form: Tablet Route of Administration: Oral
  Arms: BIVV020 with Standard of Care (SOC) Cohort A
Drug: Corticosteroids — Pharmaceutical Form: Vary Route of Administration: Vary
  Arms: BIVV020 with Standard of Care (SOC) Cohort B; Standard of Care (SOC) Cohort B

SUMMARY:
Primary Objectives:

* Cohort A: To evaluate the efficacy of BIVV020 in prevention of AMR
* Cohort B: To evaluate the efficacy of BIVV020 in treatment of active AMR

Secondary Objectives:

* To assess the overall efficacy of BIVV020 in prevention or treatment of AMR
* To characterize the safety and tolerability of BIVV020 in kidney transplant participants
* To characterize the pharmacokinetic (PK) profile of BIVV020 in kidney transplant participants
* To evaluate the immunogenicity of BIVV020

DETAILED DESCRIPTION:
Up to approximately 2 years

ELIGIBILITY:
Inclusion Criteria:

-Participant intended to receive SOC therapy per Investigator's judgment and local practice.

Cohort A: Participants with chronic kidney disease who will receive a kidney transplant from a living or deceased donor.

Cohort B: Participants who are kidney transplant recipients diagnosed with active AMR.

* BMI ≤ 40 kg/m2.
* Contraceptive use by women during the treatment period, and for at least 49 weeks after the last administration of IMP (BIVV020 + SOC arm participant) or last treatment period visit (SOC arm participant).
* Contraceptive use by men during the treatment period, and for at least 49 weeks after the last administration of IMP (BIVV020 + SOC arm participant) or last treatment period visit (SOC arm participant).

Exclusion Criteria:

* Participants who are ABO incompatible with their donors.
* Participants with known active ongoing infection as per below:

  1. Positive HIV.
  2. Positive HBV.
  3. HCV with detectable HCV RNA.
  4. Within 4 weeks of first study intervention: any serious infection, or any active bacterial infection, or any other infection which is clinically significant in the option of the Investigator, unless it can be confirmed that infection was cleared at least 3 days prior to first study intervention.
* History of active tuberculosis (TB) regardless of treatment.
* Participants with clinical diagnosis of systemic lupus erythematosus (SLE).
* Prior treatment with complement system inhibitor within 5 times the half-life.
* Current enrollment in any other clinical study where the last investigational study treatment administration was within 5 half-lives from study intervention initiation.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2026-10-26 (Estimated)

PRIMARY OUTCOMES:
Cohort A: Treatment failure rate | Up to Week 49
  Defined as the proportion of participants meeting at least one of the following criteria:
  * Biopsy-proven active AMR as per Banff Criteria 2019 as per central pathology assessment,
  * Graft loss.
Cohort B: AMR resolution rate | Up to Week 49
  Defined as the proportion of participants with post-treatment biopsy not fulfilling active AMR diagnosis criteria as per Banff Criteria 2019 as per central pathology assessment.

SECONDARY OUTCOMES:
Cohort A: Treatment failure rate per local assessment using Banff criteria 2019 | Up to Week 49
Cohort B: AMR resolution rate per local assessment using Banff criteria 2019 | Up to Week 49
Change in renal function from baseline per central laboratory assessment of estimated glomerular filtration rate (eGFR) from serum creatinine using Modification of Diet in Renal Disease equation (MDRD) | Up to 22 weeks after end of treatment period
Change in renal function from baseline per central laboratory assessment using protein: creatinine ratio | Up to 22 weeks after end of treatment period
Change in allograft histopathology Banff score | Up to Week 49
Graft survival as predicted by iBOX | Up to Week 49
Assessment of adverse events (AEs) | Up to end of study, up to approximately 2 years
  Number of participants with treatment emergent adverse events (TEAEs)/ serious adverse events (SAES), laboratory abnormalities
Change in systemic lupus erythematosus (SLE) panel | Up to 22 weeks after end of treatment period
Plasma exposure of BIVV020 assessing pharmacokinetic parameter Cmin | Up to 22 weeks after end of treatment period
  Cmin is defined as the minimum concentration after injection
Plasma exposure of BIVV020 assessing pharmacokinetic parameter AUC | Up to 22 weeks after end of treatment period
  AUC is defined as the area under plasma concentration versus time curve
Number of participants with anti-BIVV020 antibodies | Up to 22 weeks after end of treatment period
  Number of participants developed drug-induced ADAs

CONTACTS AND LOCATIONS:
Locations (27):
- United States (7):
  - Cedars-Sinai Medical Center- Site Number : 8400100, Los Angeles, California
  - University of California Los Angeles Medical Center- Site Number : 8400103, Los Angeles, California
  - University of California San Francisco - Parnassus Heights- Site Number : 8400001, San Francisco, California
  - Massachusetts General Hospital- Site Number : 8400007, Boston, Massachusetts
  - Brigham & Women's Hospital- Site Number : 8400004, Boston, Massachusetts
  - NYU Langone Medical Center- Site Number : 8400102, New York, New York
  - University of Wisconsin Hospitals and Clinics- Site Number : 8400003, Madison, Wisconsin
- Canada (4):
  - Investigational Site Number : 1240101, Vancouver, British Columbia
  - Investigational Site Number : 1240001, Vancouver, British Columbia
  - Investigational Site Number : 1240002, London, Ontario
  - Investigational Site Number : 1240003, Montreal, Quebec
- France (4):
  - Investigational Site Number : 2500007, Bordeaux
  - Investigational Site Number : 2500002, Créteil
  - Investigational Site Number : 2500001, Paris
  - Investigational Site Number : 2500005, Toulouse
- Germany (3):
  - Investigational Site Number : 2760002, Berlin
  - Investigational Site Number : 2760004, Essen
  - Investigational Site Number : 2760001, Munich
- Italy (4):
  - Investigational Site Number : 3800004, Bologna, Emilia-Romagna
  - Investigational Site Number : 3800002, Rome, Lazio
  - Investigational Site Number : 3800001, Brescia, Lombardy
  - Investigational Site Number : 3800003, Milan, Milano
- Spain (3):
  - Investigational Site Number : 7240004, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240003, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240002, Madrid, Madrid, Comunidad de
- Sweden (2):
  - Investigational Site Number : 7520001, Huddinge
  - Investigational Site Number : 7520002, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Karpman D, Bekassy Z, Grunenwald A, Roumenina LT. A role for complement blockade in kidney transplantation. Cell Mol Immunol. 2022 Jul;19(7):755-757. doi: 10.1038/s41423-022-00854-5. Epub 2022 Mar 24. No abstract available. PMID 35332298
- See also: ACT17012 kidney transplant - antibody-mediated rejection website — http://www.sanofistudies.com/O9BR/
- See also: ACT17012 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25208&tenant=MT_SNY_9011